CLINICAL TRIAL: NCT06060249
Title: Investigation of the Genetic Diseases in Infants With Unknown Cause of Death
Acronym: SIDS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, HATICE MUTLU, Assoc Prof, MD, Ankara University
Other Study IDs: SIDS2023
Record Dates: First submitted 2023-09-23; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Sudden Infant Death
MeSH Terms: conditions — Sudden Infant Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sudden infant death syndrome (SIDS) is a disease of an infant under one year of age, whose sudden death occurred unexpectedly, which the cause of death cannot be determined despite macro-autopsy, and toxicological, pathological and microbiological examinations. It is most common in babies aged 2-4 months. Although it cannot be attributed to a single cause, it is suggested that apnea/airway obstruction, abuse, developmental disorders, exposure to cigarette smoke, infections, toxic gases, metabolic diseases, and cardiac problems cause SIDS. It is known that genetic studies on SIDS are few and the literature reported so far is insufficient. On the other hand, as a result of rapid developments in genetic diagnosis methods, various genes associated with SIDS have been reported in recent studies. Most of the studies conducted include genetic studies aimed at investigating specific disease groups in SIDS. Although there are few studies on comprehensive investigation of genetic causes, potentially causative variants have been identified in 20% of cases where whole exome sequencing has been performed. In a study including perinatal deaths in which the reports of the Forensic Medicine Institute in our country were examined, 4% of the cases were reported as infant deaths of unknown cause. However, this study is only autopsy data and does not include metabolic and genetic examinations. For this reason, as far as we know, there is no information about the incidence of SIDS in our country.

Based on this information, in our research, in the province of Ankara, the deaths of children under one year of age who died unexpectedly and suddenly were examined, autopsied, and toxicological examinations were performed on internal organ samples and body fluids taken during the autopsy by the Ankara Group Presidency of the Forensic Medicine Institute between 2018 and 2023. Genetic investigation of hereditary diseases that may lead to death of cases whose cause of death cannot be explained despite pathological and microbiological examinations will be carried out by the Whole Exome Sequencing (WES) method.

The project will be carried out by researchers at Ankara University Faculty of Medicine and Forensic Medicine Institute Ankara Group Presidency. This research project was planned as a prospective, descriptive, open uncontrolled study. The duration of the project is foreseen as 12 months. Approval for our research was received from Ankara University

ELIGIBILITY:
Inclusion Criteria:

* Under one year of age, who died unexpectedly and suddenly, whose cause of death could not be determined despite the death examination, autopsy, toxicological, pathological and microbiological examinations carried out on the internal organ samples and body fluids taken during the autopsy by the Forensic Medicine Institute Ankara Group Presidency between 2018 and 2023.
* Witness blood samples taken during the autopsies of the patients will be evaluated, and peripheral blood samples of 100 patients, stored under appropriate conditions, will be transferred to the genetic laboratory for DNA isolation and genetic study.

Exclusion Criteria:

* Patients with findings indicating congenital structural anomalies or known genetic syndromes during autopsy will not be included in the study.

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This research project was planned as a prospective, descriptive, open uncontrolled study. The duration of the project is foreseen as 12 months. Approval for our research was received from Ankara University Human Research Ethics Committee.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetic diseases have an important place among the causes of sudden infant death syndrome | 1-2 years
  if a preventable cause of hereditary death is found, the families of children whose genetic cause or causes are determined are informed about the genetic disease or diseases detected, in order to prevent the occurrence of these diseases in the next pregnancy or in future generations or relatives

SECONDARY OUTCOMES:
Genetic diseases have an important place among the causes of sudden infant death | 5-10 years
  To lead the initiation of studies to detect undetected cases, to contribute to the decrease in the mortality rate of infants under one year of age (Infant mortality rate) and the mortality rate of under 5 years of age, which indicate the level of development of a country's child health and child health services, and to lead the development of preventive services for child health in our country

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice Mutlu, Ankara, Not US Or Canada, Turkey (Türkiye)